CLINICAL TRIAL: NCT06878807
Title: Eye Movements and the Extinction Procedure in Eyeblink Conditioning: A Possible Mechanism of Action for Eye Movement Desensitization and Reprocessing
Brief Title: Exploring the Role of Working Memory Saturation in Eye Movement Desensitization and Reprocessing (EMDR) Using the Eye Blink Conditioning Paradigm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Hugo López-Pelayo, Interim Junior Group Leader, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HCB/2021/0283
Record Dates: First submitted 2025-02-06; First posted 2025-03-17 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Eye Movement Desensitization and Reprocessing
MeSH Terms: interventions — Eye Movements

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Eye Movement Intervention (Experimental): Participants underwent EM tasks during the first 30 seconds of the extinction phase. All participants in this group experienced identical EM conditions in terms of speed and duration
  Interventions: Behavioral: eye movement
- TMT-B (Active Comparator): Participants performed the Trail Making Test B (TMT-B).
  Interventions: Behavioral: TMT-B
- Control group (No Intervention): Participants engaged in no additional task. These subjects were told to focus their gaze on a wall in front of them.

INTERVENTIONS:
Behavioral: eye movement — Participants underwent EM tasks during the first 30 seconds of the extinction phase. All participants in this group experienced identical EM conditions in terms of speed and duration.
  Arms: Eye Movement Intervention
Behavioral: TMT-B — Participants performed the Trail Making Test B (TMT-B).
  Arms: TMT-B

SUMMARY:
Eye Movement Desensitization and Reprocessing (EMDR) is a well-established, evidence-based treatment for posttraumatic stress disorder (PTSD). It is endorsed by leading organizations such as the American Psychiatric Association and the World Health Organization. During EMDR therapy, patients focus on recalling traumatic events while simultaneously engaging with an external stimulus. Specifically, patients undergo lateral eye movements. This process is believed to reduce the vividness and emotional intensity of traumatic memories by addressing and desensitizing their cognitive, emotional, and physical components. Despite its proven efficacy in treating PTSD, the precise mechanisms underlying these therapeutic effects remain not fully understood.

Several hypotheses have been proposed to explain the efficacy of EMDR. Among them, the working memory hypothesis is particularly influential and is supported by a substantial body of research. This hypothesis suggests that aversive memories and fear, when recalled, occupy limited memory resources. Therefore, performing a task, such as eye movements, during the recall of the traumatic experience would result in a competition for limited memory resources, leading to a decrease in the vividness and emotional intensity of the traumatic memory. Consequently, the dual task inherent in EMDR is thought to facilitate a rapid elimination of the emotional responses triggered by the traumatic memory, allowing patients to alleviate the physical and psychological distress associated with the trauma.

Measuring the effects of an EM intervention through a standardized protocol could clarify the conditions under which the intervention is most effective and elucidate the potential mechanisms of EMDR. In this context, the Eye Blink Conditioning (EBC) task, a well-established and standardized conditioning paradigm, seems relevant for testing the working memory hypothesis.

In the EBC task, eyelid closure is measured in response to a corneal air puff, which acts as the unconditioned stimulus. The unconditioned stimulus is paired with a neutral stimulus, a tone, which becomes a conditioned stimulus by eliciting a conditioned response similar to that produced by the unconditioned stimulus. After the conditioning phase, participants undergo the extinction phase. In this phase, the conditioned stimulus is presented without the unconditioned stimulus for many trials, and the main objective is to measure how many trials it takes for the participants to eliminate the previous associative learning between the aversive stimulus (air puff) and the conditioned stimulus (tone).

This study aimed to explore whether the effectiveness of a straightforward eye movement intervention in accelerating extinction is influenced by the working memory hypothesis. The hypothesis is that the enhancement of extinction learning is dependent on working memory saturation. Understanding the role of working memory saturation in the effectiveness of eye movements during extinction learning could provide critical insights into the working memory hypothesis as a potential key mechanism underlying the efficacy of EMDR therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Provide informed consent

Exclusion Criteria:

* Prior exposure to EMDR therapy or eye movement (EM) experiments
* Positive diagnosis of PTSD or other Axis I disorders as determined by the Mini-International Neuropsychiatric Interview (MINI)
* Hearing or visual impairments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Extinction Learning Differences | Baseline
  Assesses the number of conditioned responses (CR) during the initial block of the extinction phase.

SECONDARY OUTCOMES:
Latency of Eyeblink Conditioned Response (CR) During the Eye Blink Conditioning Task | Baseline
  Latency assesses the time of onset of the CR following the conditioned stimulus (CS). Data will be reported as the mean CR onset time per block.
Intensity of Eyelid Closure During the Eye Blink Conditioning Task | Baseline
  Intensity assesses the peak amplitude of the CR during conditioning trials. Data will be reported as the mean CR peak amplitude per block.
Trauma History (Childhood Trauma Questionnaire) | Baseline
  - Childhood Trauma Questionnaire (CTQ): Assesses childhood traumatic exposure. Higher scores indicate greater traumatic exposure.
Trauma History (Life Events Checklist-5) | Baseline
  - Life Events Checklist for DSM-5 (LEC-5): Evaluates exposure to 15 different types of traumatic experiences. Responses indicate whether the participant has experienced each event (Yes/No).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No